CLINICAL TRIAL: NCT06372106
Title: Philips FAST picoSAT Convenience Sampling for Clinical Performance in Neonate, Infant, and Pediatric Patients
Brief Title: Project Mountain - Comparing SpO2 and SaO2 for Accuracy
Status: Recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: MA_PM_Mountain_2022_11496
Record Dates: First submitted 2024-03-29; First posted 2024-04-17 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: SpO2; Nasal Alar Collapse, Bilateral; Oxygen; Measurement
MeSH Terms: conditions — Nasal Alar Collapse, Bilateral

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Neonates: Even distribution of sex per skin pigmentation category (Light, Medium, Dark)
  Interventions: Device: SaO2 Sampling
- Infants: Even distribution of sex per skin pigmentation category (Light, Medium, Dark)
  Interventions: Device: SaO2 Sampling
- Pediatrics: Even distribution of sex per skin pigmentation category (Light, Medium, Dark)
  Interventions: Device: SaO2 Sampling

INTERVENTIONS:
Device: SaO2 Sampling — CO-Oximetry analysis of arterial blood samples

SUMMARY:
The main goal of this study is to look at the performance of the neonatal, infant, and pediatric Philips SpO2 sensors with the Philips FAST Pulse Oximetry technology. Oxygen saturation measurements (SpO2) will be obtained via pulse oximetry and invasive arterial oxygen measurements (SaO2) will be obtained via arterial blood samples as part of your clinical care and assessed by co-oximetry. The study will aim to enroll a diverse population to help us understand the impact of skin pigmentation.

DETAILED DESCRIPTION:
This is a prospective, multi-center, multi-phase, unblinded, non-randomized. self-controlled, observational study. All data analyses specified below will be calculated and summarized by each of SpO2 sensors under test. Demographics and baseline characteristics, including sex assigned at birth, age, ethnicity, race, baseline height, baseline weight, BMI, skin pigmentation and sensor application site measurements will be summarized with descriptive statistics using the analysis set.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 years or older or parent/legal guardian of subject aged less than 18 years, willing and able to understand and provide written informed consent/assent.
* Weight and/or age within intended use of at least one SpO2 sensor under test at time of enrollment.
* Willing and able to wear study devices in addition to SoC devices and during SoC procedures.
* In-patient within a neonatal or pediatric intensive care unit (e.g. NICU, PICU, PCICU).
* Has arterial access and ability to have arterial blood samples drawn as part of their SoC and analyzed by CO-Oximetry.

Exclusion Criteria:

* Known pregnancy or lactating females (self-reported)
* Injury, wounds, physical malformation, hyperkeratosis, or compromised/non-intact skin at sensor application site (i.e. fingers, toes, hands, feet, ears, nasal ala). Note: Certain malformations may be allowed if determined it would not affect application of sensor with the pulse oximetry system.
* Self-reported severe contact allergies to standard adhesives or other materials found in pulse oximetry sensors. Note: Subject may be considered eligible if subject can wear non-adhesive sensor.
* Unwillingness or inability to remove nail polish or artificial nails from sensor application site.
* Nail fungus on sensor application site.
* Wearing and unable to remove jewelry from sensor application site.
* Dye injection within 48 hours of enrollment.
* Known dysfunctional hemoglobin levels (COHb >3%, MetHb >2%, and ctHb <10g/dl)
* Undergoing phototherapy for neonatal hyperbilirubinemia during arterial blood sampling

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted in neonate, infant, and pediatric patients admitted into an intensive care unit (e.g. NICU, PICU, PCICU).
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To observed accuracy expressed in ARMS of SpO2 measurements obtained from neonatal, infant, and pediatric sensors with the Philips FAST Pulse Oximetry technology within the range of 70-100% in comparison to the SaO2 as ground truth. | through study completion, an average of 8 months
  The oximetry technology will be expressed in ARMS of SpO2 measurements obtained from neonatal, infant, and pediatric sensors with the Philips FAST Pulse Oximetry technology within the range of 70-100% in comparison to the SaO2 as ground truth.

SECONDARY OUTCOMES:
Secondary Endpoint -Non-disparate bias with consideration to skin pigmentation for each neonatal, infant, and pediatric SpO2 sensor under test with the Philips FAST Pulse Oximetry technology. | through study completion, an average of 8 months
  Non-disparate bias with consideration to skin pigmentation for each neonatal, infant, and pediatric SpO2 sensor under test with the Philips FAST Pulse Oximetry technology.
Secondary Endpoint- Proportion of paired SaO2 and SpO2 readings in which occult hypoxemia (i.e., SaO2 <88% with SpO2 ≥92%) is identified among patients within the broad categories of light, medium, and dark pigmentation. | through study completion, an average of 8 months
  Proportion of paired SaO2 and SpO2 readings in which occult hypoxemia (i.e., SaO2 <88% with SpO2 ≥92%) is identified among patients within the broad categories of light, medium, and dark pigmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Azer, Study Director — Philips Healthcare
Locations (5):
- United States (5):
  - Phoenix Children's, Phoenix, Arizona
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No